CLINICAL TRIAL: NCT05910710
Title: Impact of Immuno-Oncologic Agent on Neoadjuvant Chemotherapy in Triple Negative Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Other Study IDs: 2023-02-019
Record Dates: First submitted 2023-06-06; First posted 2023-06-20 (Actual); Last update posted 2023-06-20 (Actual); Status verified 2023-06

CONDITIONS: Triple Negative Breast Cancer; Neoadjuvant Chemotherapy; Pembrolizumab; Tumor Microenvironment
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Biospecimen Retention: Samples With DNA — Blood : Germline DNA Tissue : DNA/RNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Subjects administered Neoadjuvant Pembrolizumab: Neoadjuvant Weekly paclitaxel, Carboplatin followed by Doxorubicin, Cyclophosphamide add Pembrolizumab
  Interventions: Genetic: Visium, Whole Genome Sequencing(WGS)/Whole Transcriptome Sequencing(WTS)
- Subjects not administered Neoadjuvant Pembrolizumab: Neoadjuvant Weekly paclitaxel, Carboplatin followed by Doxorubicin, Cyclophosphamide
  Interventions: Genetic: Visium, Whole Genome Sequencing(WGS)/Whole Transcriptome Sequencing(WTS)

INTERVENTIONS:
Genetic: Visium, Whole Genome Sequencing(WGS)/Whole Transcriptome Sequencing(WTS) — Visium : Spatial transcriptomics WGS/WTS : detection of somatic mutation

SUMMARY:
It analyzes the Tumor microenvironment(TME) changes in non pathologic complete response(pCR) subjects among subjects who were administered neoadjuvant pembrolizumab and those who were not administered neoadjuvant pembrolizumab for triple negative breast cancer.

(Neoadjuvant Weekly paclitaxel, Carboplatin +- Pembrolizumab followed by Doxorubicin, Cyclophosphamide +- Pembrolizumab regimen)

ELIGIBILITY:
Inclusion Criteria:

* Triple negative breast cancer
* Subjects administered neoadjuvant Weekly paclitaxel, Carboplatin followed by Doxorubicin, Cyclophosphamide add Pembrolizumab or not
* Non pCR patients who are undergoing surgery after neoadjuvant chemotherapy
* Sign to informed consent

Exclusion Criteria:

* Patients with difficulty in obtaining sufficient samples

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally advanced triple negative breast cancer subjects who were administered neoadjuvant chemotherapy with Weekly paclitaxel, Carboplatin followed by Doxorubicin, Cyclophosphamide add Pembrolizumab or not
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-03-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Genomic profiling will be assessed by tissue and blood samples(analyze the TME changes) | 3year
  Tissue and blood will be tested for Spatial transcriptomics, WGS(Wilcoxon rank sum test or Chi-square test, cell-cell interaction)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea